CLINICAL TRIAL: NCT00241111
Title: Assessment of the Efficacy, Tolerability and Pharmaco-economic Impact of Zoledronic Acid Treatment in Prostate Cancer With Bone Metastasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EFR04
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2010-04

CONDITIONS: Prostate Cancer With Bone Metastasis
Keywords: Prostate; cancer; bone metastasis; zoledronic acid
MeSH Terms: conditions — Neoplasms | interventions — Zoledronic Acid

ARMS (1):
- Zometa (Other)
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: zoledronic acid
  Other Names: ZOl446

SUMMARY:
Study to determine effectiveness and safety of zoledronic acid and whether it has a pharmaco-economic impact in prostate cancer with bone metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years.
* Written informed consent.
* With histologically-proven prostate carcinoma.
* ECOG performance status ≤ 2
* Life expectancy > 12 months
* Current or previously documented diagnosis of at least 1 bone metastasis due to prostate cancer (patient could be hormono naif, Hormono sensible or hormono refractory)
* Patients with partners of childbearing potential should use a barrier method of contraception throughout the study.

Exclusion Criteria:

* ECOG performans status >3
* Prior treatment with bisphosphonates IV within the last 3 month to the study
* Renal insufficiency (serum creatinine > 265 micromol/L or > 3.0 mg/dL)
* Liver function tests > 2.5 ULN
* Patients with another nonmalignant disease which would confuse the evaluation of primary endpoints or prevent the patient from complying with the protocol.
* History of concomitant disease with influence on bone metabolism such as Paget's disease or primary hyperparathyroidism
* Disabling or non controlled concomitant disease likely to alter the quality of life
* Patient unable to fill in a questionnaire: senile dementia, psychiatric or neurological disease, illiterate or partially sighted patient
* Known hypersensitivity to zoledronic acid or other bisphosphonates

Other protocol-defined inclusion / exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2003-09; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
to assess the effectiveness of Zol in prevention of SREs in stratified groups (hormonal treatment) | at 15 months & at end of study

SECONDARY OUTCOMES:
to assess the effectiveness of Zol in improving pain and QoL in prostate cancer patients with bone metastases | V1, V2, V3, V5
to assess the safety of ZOL treatment | V1, V2, V3, V5
to assess resources consumption | V1, V2, V3, V5
to assess BM | V1 et V5

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals